CLINICAL TRIAL: NCT02100072
Title: Evaluation of 1440nm Laser Assisted Selective Photothermolysis for Treatment of Axillary Hyperhidrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cynosure, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CYN13-MK-HH01
Record Dates: First submitted 2014-03-25; First posted 2014-03-31 (Estimated); Results first posted 2020-12-11 (Actual); Last update posted 2021-01-08 (Actual); Status verified 2020-12

CONDITIONS: Hyperhidrosis
MeSH Terms: conditions — Hyperhidrosis | interventions — Lasers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nd:YAG 1440 nm laser (Experimental)
  Interventions: Device: Nd:YAG 1440 nm laser

INTERVENTIONS:
Device: Nd:YAG 1440 nm laser

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of the Nd:YAG 1440 nm wavelength laser for the treatment of primary hyperhidrosis of the axilla.

ELIGIBILITY:
Inclusion Criteria:

* A healthy non-smoking male or female between 18-55 years of age
* Understand/accept obligation not to receive any other procedures in anatomical areas exhibiting axillary hyperhidrosis through 3 months prior to treatment
* Understand and accept the obligation and is logistically able to present for all scheduled follow-up visits
* Clinically diagnosed for primary hyperhidrosis of the axilla.
* A self-assessed Hyperhidrosis Disease Severity Scale (HDSS) score of three (3) or four (4)

Exclusion Criteria:

* Clinical diagnosis of secondary hyperhidrosis
* Uncontrolled systemic disease or infection
* Concurrent use of any hyperhidrosis treatments other than over the counter antiperspirants or deodorants
* Receipt of Botox® or Dysport® within the past six months
* Patients who refuse to stop using over the counter antiperspirants 24 hours prior to the day of surgery and each of the follow-up visits at 3 months and 6 months that Minors starch iodine tests may be performed.
* Patients using or having used within 7 days of baseline visit: cholinomimetic agents, anticholinergic agents, prescription antiperspirants, any herbal medicine treatments or any other treatments for hyperhidrosis except over the counter antiperspirant or planning to use such agents during the course of the study.
* Any previous liposuction/liposculpture or any type of surgery for hyperhidrosis; OR any other types of treatments for hyperhidrosis in the area to be treated in the past 6 months
* Has any other medical condition, that, in the investigator's opinion would interfere with the subject's participation in the study
* Is susceptible to light induced seizures or history of seizures
* Has a history of keloid formation
* Significant cardiovascular disease
* Bleeding disorders
* Anti-platelet and anticoagulant medication
* Sensitivity to lidocaine or epinephrine
* Pregnancy or planned pregnancy
* Existing neuromuscular disorders (myasthenia gravis, Eaton-Lambert Syndrome, amyotrophic lateral sclerosis)
* Electronic implants
* Subjects requiring supplemental oxygen
* Has therapies or medications which may interfere with the treatment (including medications causing photosensitivity
* Allergic to Doxycycline

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2013-06; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Krantz, Study Director — Cynosure, Inc.
Locations (1):
- Skin Care Physicians, Chestnut Hill, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Nd:YAG 1440 nm Laser: Nd:YAG Laser With 1440nm Wavelength.
  Each subject received 1 treatment using this laser over an approximately 3x4 cm area.
Period: Overall Study
Arm/Group | Nd:YAG 1440 nm Laser
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Nd:YAG 1440 nm Laser: Nd:YAG 1440 nm laser
Arm/Group | Nd:YAG 1440 nm Laser
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Caucasian | 3
  Race/Ethnicity: African American | 2
Fitzpatrick Skin Score [Count of Participants; unit: Participants] — The Fitzpatrick Skin Score is used to determine skin color. It is a numerical system that classifies skin into six types (Type I, Type II, Type III, Type IV, Type V and Type VI) based on the numerical score achieved (ranging from 0 to 36). The lower the score (and skin type number), the fairer the skin. The higher the score (and skin type number), the more deeply pigmented the skin is.
  The scale comes from this source:
  Gupta, Sharma. Skin typing: Fitzpatrick grading and others. Clinics in Dermatology. 2019;37(5):430-436. doi:10.1016/j.clindermatol.2019.07.010
  Participants
    Fitzpatrick Skin Type I | 0
    Fitzpatrick Skin Type II | 0
    Fitzpatrick Skin Type III | 3
    Fitzpatrick Skin Type IV | 0
    Fitzpatrick Skin Type V | 2
    Fitzpatrick Skin Type VI | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Sweating Assessed Using Gravimetry
Description: A gravimetry test was performed to determine the quantity of sweat produced, comparing the post-treatment to the baseline numbers. A pre-weighted filter paper was placed on the armpit, and then weighed afterwards to determine the quantity of sweat produced. To calculate the change between the baseline and 3 months post baselines, the values taken at these 2 time points are subtracted from each other. A negative value means that there has been a decrease in gravimetric weight since the baseline.
Time Frame: Baseline and 3 months post baseline
Population: 1 subject was incapable of attending the follow up visit, so their gravimetric measurement was not able to be obtained. They were able to answer other follow up questions via the phone, however.
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Nd:YAG 1440 nm Laser
Number analyzed (Participants) | 4
mg
  Average Gravimetric Change (Left Side) | -104.50 (156.57)
  Average Gravimetric Change (Right Side) | -90.85 (131.84)

ADVERSE EVENTS:
Time Frame: Adverse Events occurring were captured and followed throughout the study duration, approximately 3 months.
Arm/Group | Nd:YAG 1440 nm Laser
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 2/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nd:YAG 1440 nm Laser (N=5)
Sweat (Skin and subcutaneous tissue disorders) | 1
Numbness (Nervous system disorders) | 2
Bruising (Skin and subcutaneous tissue disorders) | 1
Itching (Skin and subcutaneous tissue disorders) | 1
Pain (Nervous system disorders) | 2
Redness (Skin and subcutaneous tissue disorders) | 1
Swelling (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI cannot disclose confidential or proprietary information until after it becomes generally known or available to the public.